CLINICAL TRIAL: NCT05197699
Title: A Multicenter, Prospective Cohort Study to Document the Immunization Status of MS Patients in Germany With Focus on Anti-SARS-CoV-2 Vaccination Response
Brief Title: Severe Acute Respiratory Syndrome Coronavirus Type 2 (SARS-CoV-2)-Related Multiple Sclerosis (MS) Vaccination Study
Status: Terminated | Type: Observational
Why Stopped: Sponsor's decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: DE-MSG-11922
Record Dates: First submitted 2022-01-17; First posted 2022-01-19 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis (MS)
Keywords: SARS-Cov2 vaccination
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DMT-Treated Participants: MS participants who are receiving DMTs will be enrolled.
- Untreated Participants: MS participants who are receiving no DMT treatment or receiving only symptomatic treatment will be enrolled.

SUMMARY:
The primary objective of this study is to document immunization status of MS participants after SARS-CoV-2-vaccinations and to evaluate possible effects of disease modifying therapy (DMTs) on the immune status. The secondary objectives of the study are to document longevity of immunization status of MS participants after SARS-Cov-2-vaccinations and to evaluate possible effects of DMTs on the immune status, to assess anti SARS-CoV-2 antibody titers regarding amount and persistence, to document immunization status of MS participants after repeated SARS-Cov-2-vaccinations and to evaluate possible effects of DMTs on the immune status, to document vaccine types used in MS population in Germany and to describe tolerability of SARS-CoV-2 vaccines according to participant's assessment.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of MS according to McDonald criteria (2018)
* SARS-CoV-2 vaccination is planned (within the upcoming 90 days), underway (only one of two vaccinations received) or only recently completed (in the last 6 weeks) or SARS-CoV-2 vaccination has been completed >6 weeks but an additional vaccination is planned within the upcoming 30 days

Key Exclusion Criteria:

* Participant cannot be regularly followed up for organizational or geographic reasons
* Participant is unwilling to get vaccinated against SARS CoV-2 virus

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are receiving any type of DMTs and participants who do not receive any medicinal treatment for their MS or receive only symptomatic treatment will be enrolled.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Developed an Immune Response to Their Last SARS-CoV-2-Vaccination | 30 days after the last vaccination

SECONDARY OUTCOMES:
Number of Participants who Retained an Immune Response to Their Last SARS-CoV-2-Vaccination | 6 months after 2nd vaccination
Change From Baseline in SARS-CoV-2 Spike Immunoglobulin A (IgA) Levels | Baseline up to 6 months after 2nd vaccination
Change From Baseline in SARS-CoV-2 Spike Immunoglobulin G (IgG) Levels | Baseline up to 6 months after 2nd vaccination
Change From Baseline in SARS-CoV-2-Nucleocapsid Protein (NCP) IgG Levels | Baseline up to 6 months after 2nd vaccination
Number of Participants who Developed an Immune Response to Their SARS-CoV-2-Vaccination | 28 days after 2nd vaccination and 6 months after 2nd vaccination
Number of Participants by Applied SARS-CoV-2 Vaccine and Vaccination Cycle | Up to 33 months
Number of Participants per Vaccination Cycle | Up to 33 months
Number of Participants with the Tolerability to the Applied Vaccine According to the Predefined Categories | Up to 33 months
  Predefined categories for assessing tolerability are tolerated better than expected, as expected, and worse than expected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (12):
- Germany (12):
  - Multiple Sklerose Zentrum, Bamberg
  - St. Josef Hospital, Klinikum der Ruhr-Universität Bochum, Bochum
  - Universitätsklinikum Erlangen, Neurologische Klinik, Erlangen
  - Universitätsklinik Freiburg, Neurologie, Freiburg im Breisgau
  - Klinik für Neurologie, Haar
  - UKE Hamburg, Klinik und Poliklinik für Neurologie, Hamburg
  - Univ.-Klinikum Heidelberg, Neurologische Klinik, Heidelberg
  - Klinik und Poliklinik für Neurologie, Leipzig
  - Klinik und Poliklinik für Neurologie, Munich
  - Universitätsklinikum Tübingen, Neurologie, Tübingen
  - Neuropraxis München Süd, Unterhaching
  - DKD Helios Klinik, Neurologie, Wiesbaden

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/